CLINICAL TRIAL: NCT04880954
Title: Soft Tissue Mobilization and Rehabilitation on Pain and Physical Functioning for Non-Specific Chronic Knee Pain: A Randomized Clinical Trail
Brief Title: Manual Therapy and Rehabilitation on Pain and Physical Functioning for Chronic Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuro Performance Integration (Other)
Responsible Party: Principal Investigator, Beverly Albert, Research Director, Neuro Performance Integration
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #21-NPI-101
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Non-Specific Chronic Knee Pain
MeSH Terms: interventions — Musculoskeletal Manipulations; Rehabilitation; Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups 1) Manual Therapy, 2) Rehabilitation, or 3) Combination of both
Masking Description: Participants will know the group they are randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soft Tissue Mobilization (Experimental)
  Interventions: Procedure: Soft Tissue Mobilization
- Rehabilitation (Experimental)
  Interventions: Other: Rehabilitation
- Soft Tissue Mobilization and Rehabiliation (Experimental)
  Interventions: Procedure: Soft Tissue Mobilization; Other: Rehabilitation

INTERVENTIONS:
Procedure: Soft Tissue Mobilization — Soft Tissue Mobilization will be provided to participants by Licensed Chiropractor focusing on structures of the lower and upper leg. This will be provided for 20 minutes, once per week for 12 weeks.
  Other Names: Manual Therapy
  Arms: Soft Tissue Mobilization; Soft Tissue Mobilization and Rehabiliation
Other: Rehabilitation — Participants will engage in 20 minutes of prescribed at-home exercise 5 times per week, for 12 weeks.
  Other Names: Injury Prevention Therapy; Isometric Exercise
  Arms: Rehabilitation; Soft Tissue Mobilization and Rehabiliation

SUMMARY:
This is a research study examining if hands-on therapy and prescribed exercise is an effective way to manage and reduce knee pain. It will also look at physical benefits of this treatment including balance, strength, and flexibility.

Participation will include 2 assessment days and a 12-week treatment cycle. Assessments will be conducted during week 1 and after treatment. The treatment will vary based on the assigned group. This may include 12 in-person manual therapy sessions occurring once per week and or 12-weeks of at-home therapy occurring 5 times per week.

The greatest risk of participation includes possible muscle/joint soreness, injury during at-home exercises, and loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Adults experiencing non-specific knee pain for 3 or more months. Pain must be 3/10 (VAS) or higher.

Exclusion Criteria:

* Pain due to knee surgery, fracture, tumor, trauma, or those on medication for mood disorder (assessed on case by case basis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Pain | This will be measured pre- and post- intervention (week 1 and week 13).
  The Visual Analogue Scale (VAS) will be used to quantify pain. The scale ranges from 1 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Range of Motion | This will be measured pre- and post- intervention (week 1 and week 13)
  A goniometer will be used to assess range of motion of the hip and knee.
Modified Clinical Test of Sensory Integration and Balance | This will be measured pre- and post- intervention (week 1 and week 13).
  The Balance Tracking System will be used to assess balance.
Isometric Strength | This will be measured pre- and post- intervention (week 1 and week 13).
  A crane scale will be used to measure changes in isometric strength (pounds). The hamstring and quadricep will be assessed.
Limits of Stability | This will be measured pre- and post- intervention (week 1 and week 13).
  The Balance Tracking System will be used to assess limits of stability.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Albert, MS, Principal Investigator — Neuro Performance Integration
Locations (1):
- Neuro Performance Integration, Park City, Utah, United States

IPD SHARING:
Plan to Share IPD: No